CLINICAL TRIAL: NCT04493840
Title: Effect of Shenfu Injection on Myocardial Injury in Patients With Acute ST Segment Elevation Myocardial Infarction After Primary Percutaneous Coronary Intervention: A Multicenter, Randomized, Double-Blinded, Parallel-Group, Placebo-Controlled Clinical Trial
Brief Title: Randomized Evaluation of Shenfu Injection to Reduce Myocardial Injury
Acronym: RESTORE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine, Director, Emergency & Critical Care Center, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019013
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Shen-Fu; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shenfu Injection (Experimental)
  Interventions: Drug: Shenfu Injection
- 5% Glucose Injection (Placebo Comparator)
  Interventions: Drug: 5% Glucose Injection

INTERVENTIONS:
Drug: Shenfu Injection — 80ml Shenfu Injection + 70ml 5% glucose injection, ivdrip, within 30 minutes before PCI and 1 to 5 days (once a day) after PCI (6 times in total). Drug titration time should be no less than 30 minutes.
  Arms: Shenfu Injection
Drug: 5% Glucose Injection — 150 ml 5% glucose injection, ivdrip, within 30 minutes before PCI and 1 to 5 days (once a day) after PCI (6 times in total). Drug titration time should be no less than 30 minutes.
  Arms: 5% Glucose Injection

SUMMARY:
This study aims to evaluate whether perioperative use of Shenfu Injection, as compared to placebo, could reduce infarct size assessed by cardiac magnetic resonance (CMR) in patients with acute anterior ST-segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Shenfu injection is a traditional Chinese medicine formulation containing ginseng (Panax; family: Araliaceae) and aconite (Radix aconiti lateralis preparata, Aconitum carmichaeli Debx; family: Ranunculaceae) with Ginsenosides and aconite alkaloids as the main active ingredients. Its quality is strictly controlled in compliance with the standard of the China Ministry of Public Health (official approval code: certification number Z20043117; No. 110804, Ya'an, China). Animal studies have shown that Shenfu injection has protective effects against reperfusion injury through multiple pharmacologic effects, including scavenging free radicals, inhibiting inflammatory mediators, suppressing cell apoptosis, and inhibiting calcium overload. However, few data are available regarding its efficacy in humans. We aimed to determine whether perioperative use of Shenfu injection, as compared to placebo, might reduce infarct size in patients with STEMI undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <75 years.
2. First-time acute anterior STEMI scheduled for primary PCI.
3. ST segment elevation in at least two contiguous precordial leads according to electrocardiogram (>30 min).
4. Symptoms onset ≤12 hours.
5. The presence of proximal or middle left anterior descending branch (LAD) occlusion with pre-PCI TIMI flow 0 or 1 according to baseline coronary angiogram.
6. Written informed consent.

Exclusion Criteria:

1. Cardiogenic shock, serious heart failure (Killip class III or above), malignant ventricular arrhythmia, or mechanical complications.
2. Post cardiopulmonary resuscitation (CPR) (including cardioversion).
3. Patients who have received thrombolytic therapy or upstream GPIIb/IIIa inhibitors (GPI).
4. Uncontrolled hypertension (systolic BP ≥180 mm Hg or a diastolic BP ≥110 mmHg).
5. Prior myocardial infarction, PCI or coronary artery bypass graft.
6. Known severe hepatic insufficiency (AST/ALT >3-fold the upper limit of normal value) or known renal insufficiency.
7. Malignant tumor, lymphoma, HIV-positive, or cirrhosis with life expectancy <1 year.
8. Patients with active bleeding, intracranial hemorrhage, major surgery or trauma within 1 months, or ischemic stroke or transient ischemic attack (TIA) within 6 months.
9. History of anemia (hemoglobin<90g/L) or thrombocytopenia (thrombocyte<100×109/L).
10. Patients who require simultaneous intervention of left main disease during primary PCI or those with multi-vessel disease who plan to intervene in non-culprit vessels within 7 days (simultaneous or staged).
11. Scheduled for CABG within one month after randomization.
12. Pregnancy, lactation, or potentially fertile women.
13. Patients who have known to be allergic to Shenfu Injection or its components or patients with serious adverse effect.
14. Patients with contraindication to CMR (metal foreign body in the body, claustrophobia, etc.).
15. Participation in other clinical trial in recent 3 months.
16. Patients who cannot complete this trial or comply with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Infarct size (% of left ventricular mass) | 5±2 days after PCI
  Infarct size was assessed by performing CMR imaging at 5±2 days after PCI

SECONDARY OUTCOMES:
Microvascular obstruction (% of left ventricular mass) | 5±2 days after PCI
Intramyocardial hemorrhage (% of left ventricular mass) | 5±2 days after PCI
Area under the curve (AUC) of creatine kinase isoenzyme (CK-MB) | Immediately after admission (0 hour), and 6, 12, 18, 24, 48, and 72 hours after PCI
AUC of cardiac troponin I | Immediately after admission (0 hour), and 6, 12, 18, 24, 48, and 72 hours after PCI
Peak value of CK-MB and cTnI | 72 hours after PCI
ST segment resolution (%) according to ECG | 24 hours after PCI
TIMI flow grade | Immediately after PCI
Corrected TIMI frame count (CTFC) | Immediately after PCI
TIMI myocardial perfusion grade (TMPG) | Immediately after PCI
Myocardial salvage index | 5±2 days after PCI
Area at risk (myocardial edema, % of left ventricular mass) | 5±2 days after PCI
Left ventricular end-diastolic volume (LVEDV) | 5±2 days after PCI
Left ventricular end-systolic volume (LVESV) | 5±2 days after PCI
Left ventricular ejection fraction (LVEF) | 5±2 days after PCI
Major adverse cardiovascular and cerebrovascular events (MACCE, including cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, emergency revascularization) | 30 days after PCI
Individual events (including cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, emergency revascularization, re-hospitalization for heart failure) | 30 days after PCI

OTHER OUTCOMES:
Slow flow and no flow | Index procedure
Malignant arrhythmia (ventricular fibrillation, ventricular tachycardia, etc.) | Index procedure
Value of high-sensitivity C-reactive protein (Hs-CRP) | Immediately after admission (0 hour), and 24, 72 hours and 5 days after PCI
Value of brain natriuretic peptide (BNP) | Immediately after admission (0 hour), and 24, 72 hours and 5 days after PCI
The Myocardial Infarction Dimensional Assessment Scale (MIDAS) | 6 hours and 30 days after PCI
  0 to 140 scores, higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Wang X, Guo R, Guo Y, Guo Q, Yan Y, Gong W, Zheng W, Wang H, Xu L, Ai H, Que B, Yan X, Ma X, Nie S. Rationale and design of the RESTORE trial: A multicenter, randomized, double-blinded, parallel-group, placebo-controlled trial to evaluate the effect of Shenfu injection on myocardial injury in STEMI patients after primary PCI. Am Heart J. 2023 Jun;260:9-17. doi: 10.1016/j.ahj.2023.02.005. Epub 2023 Feb 22. PMID 36822255